CLINICAL TRIAL: NCT00434213
Title: A Phase IV, Multi-center, Open-label Study of DAYTRANA (Methylphenidate Transdermal System [MTS]) to Characterize the Dermal Reactions in Pediatric Patients Aged 6-12 With Attention Deficit/Hyperactivity Disorder (ADHD).
Brief Title: Characterization of Dermal Reactions in Pediatric Patients With ADHD Using DAYTRANA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Noven Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPD485-411
Record Dates: First submitted 2007-02-12; First posted 2007-02-13 (Estimated); Results first posted 2009-03-06 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-03

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Methylphenidate Transdermal System (Experimental): To characterize the dermal reactions seen with the use of DAYTRANA
  Interventions: Drug: Daytrana

INTERVENTIONS:
Drug: Daytrana — Methylphenidate Transdermal System (MTS)
  Other Names: MTS

SUMMARY:
This is a study designed to characterize the dermal response of DAYTRANA. Subjects will visit the study site over a period of approximately 14 weeks.

DETAILED DESCRIPTION:
This is a study designed to characterize the dermal response of DAYTRANA. Subjects will visit the study site over a period of approximately 14 weeks. Subjects will be titrated to an optimum dose of study treatment and assessed for safety and efficacy. Dermal response will be evaluated at each visit by the investigator. Subjects with high dermal response scores or scores that persist at the same application site and have no improvement after up to 4 evaluations (not to exceed a two week period) will be discontinued from the study and referred to a study specific dermatologist for specialized skin sensitivity skin patch testing.

ELIGIBILITY:
Inclusion Criteria:

* Must sign informed consent.
* Male or female 6-12 years old.
* Negative pregnancy test.
* Meet Diagnostic and Statistical Manual of Mental Disorders, 4th edition - Text Revision (DSM-IV-TR) criteria for a primary diagnosis of ADHD.
* No co-morbid illness that could affect safety, tolerability or interfere with participation.
* Blood pressure (BP) within the 95th percentile for age, gender, and height.
* Willing and able to comply with all the requirements defined in protocol.

Exclusion Criteria:

* Current controlled (requiring a restricted medication) or uncontrolled co-morbid psychiatric diagnosis (except Oppositional Defiant Disorder [ODD]).
* At risk for suicidal or violent behavior towards self or others.
* History of a suicide attempt.
* History of a structural cardiac abnormality or other serious cardiac problems.
* Non-responder to psychostimulant treatment.
* Is overweight.
* Seizures during the last 2 years (exclusive of infantile febrile seizures), a tic disorder, a current diagnosis and/or family history of Tourette's Disorder.
* Has Conduct Disorder.
* Known history of alcohol or other substance abuse within the last 6 months.
* Any abnormal thyroid function.
* A concurrent chronic or acute illness, disability, or other condition that might confound results of safety assessments.
* Has had treatment with any known liver altering agents within 30 days prior to Screening.
* Taking any excluded medication.
* Previous use of DAYTRANA.
* Taking other medications that have Central Nervous System (CNS) effects.
* Female subject is pregnant or lactating.
* Has any skin disease, or history of any chronic skin disease, skin cancer, skin manifestations of allergic disease, or other dermatologic conditions.
* Has sensitive-skin syndrome or has sensitivities to the ingredients in soaps, lotions, cosmetics or adhesives.
* Has clinical signs and symptoms of skin irritation or hyper/hypopigmentation at the potential application sites.
* A documented allergy, hypersensitivity or intolerance of methylphenidate (MPH) or any components found in DAYTRANA.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 309 (Actual)
Dates: Start 2007-01; Primary Completion 2007-08 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Wilens, MD, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (29):
- United States (29):
  - Scottsdale, Arizona
  - Irvine, California
  - San Marcos, California
  - Spring Valley, California
  - Wildomar, California
  - Boulder, Colorado
  - Gainesville, Florida
  - Miami, Florida
  - Winter Park, Florida
  - Libertyville, Illinois
  - Northbrook, Illinois
  - Overland Park, Kansas
  - Bardstown, Kentucky
  - Owensboro, Kentucky
  - Cambridge, Massachusetts
  - Kalamazoo, Michigan
  - Las Vegas, Nevada
  - Toms River, New Jersey
  - Rochester, New York
  - Cleveland, Ohio
  - Columbus, Ohio
  - Portland, Oregon
  - Salem, Oregon
  - Philadelphia, Pennsylvania
  - Jackson, Tennessee
  - Austin, Texas
  - Lubbock, Texas
  - San Antonio, Texas
  - Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Warshaw EM, Squires L, Li Y, Civil R, Paller AS. Methylphenidate transdermal system: a multisite, open-label study of dermal reactions in pediatric patients diagnosed with ADHD. Prim Care Companion J Clin Psychiatry. 2010;12(6):PCC.10m00996. doi: 10.4088/PCC.10m00996pur. PMID 21494336

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Daytrana
Started | 309
Completed | 260
Not Completed | 49
Not completed — Adverse Event | 12
Not completed — Lack of Efficacy | 9
Not completed — Lost to Follow-up | 14
Not completed — Withdrawal by Subject | 7
Not completed — Protocol Violation | 3
Not completed — Unable to comply with study visit window | 2
Not completed — Application site reaction | 1
Not completed — Non-compliant to study schedule | 1

BASELINE CHARACTERISTICS:
Arm/Group | Daytrana
Number analyzed (Participants) | 309
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 309
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.1 (1.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91
  Male | 218
Region of Enrollment [Number; unit: participants]
  United States | 309

OUTCOME MEASURES:

1. Primary Outcome: Dermal Reactions
Description: Dermal reactions were graded on a scale ranging from 0 (no irritation) to 7 (strong reaction) for observed findings of erythema, edema, papules, and vesicles.
Time Frame: 7 weeks
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | Daytrana
Number analyzed (Participants) | 305
Participants
  0 (no evidence of irritation) | 46
  1 (minimal erythema) | 97
  2 (definite eythema) | 151
  3 (erythema and papules) | 6
  4 (definite edema) | 3
  5 (erythema, edema, and papules) | 0
  6 (vesicular eruption) | 0
  7 (strong reaction beyond test site) | 0
  No dermal evaluation | 2

2. Secondary Outcome: Contact Sensitization to Methylphenidate
Description: Contact sensitization to methylphenidate through skin patch testing.
Time Frame: 7 weeks
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | Daytrana
Number analyzed (Participants) | 305
Participants | 1

ADVERSE EVENTS:
Arm/Group | Daytrana
Serious Adverse Events (participants affected / at risk) | 0/305
Other Adverse Events (participants affected / at risk) | 242/305
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daytrana (N=305)
Decreased appetite (Metabolism and nutrition disorders) | 95 (99)
Headache (Nervous system disorders) | 50 (64)
Insomnia (Psychiatric disorders) | 32 (34)
Abdominal pain upper (Gastrointestinal disorders) | 26 (36)
Affect lability (Psychiatric disorders) | 22 (26)
Nausea (Gastrointestinal disorders) | 22 (27)
Upper respiratory tract infection (Infections and infestations) | 20 (20)
Irritability (Psychiatric disorders) | 18 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after SPONSOR confirms there shall be no multicenter Study publication, the INSTITUTION and/or such PRINCIPAL INVESTIGATOR may publish the results from the INSTITUTION site individually.